CLINICAL TRIAL: NCT06505681
Title: Pragmatic Randomized Controlled Trial of Pharmacopuncture Therapy for Chronic Knee Pain: A Pilot Study
Brief Title: Pharmacopuncture Therapy for Chronic Knee Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Jaseng Medical Foundation (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: JS-CT-2022-16
Record Dates: First submitted 2024-07-11; First posted 2024-07-17 (Actual); Last update posted 2024-07-17 (Actual); Status verified 2024-07

CONDITIONS: Chronic Knee Pain
Keywords: Chronic knee Pain; Pharmacopuncture
MeSH Terms: interventions — Physical Therapy Modalities

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Pharmacopuncture (Experimental): 20 patients with pharmacoacupuncture
  Interventions: Procedure: Pharmacopuncture
- Physical therapy (Active Comparator): 20 patients with physical therapy
  Interventions: Procedure: Physical therapy

INTERVENTIONS:
Procedure: Pharmacopuncture — The selection of acupoints, depth of insertion, and other parameters will be determined based on the clinical judgment of the Korean medicine practitioner, considering the patient's symptoms, imaging results, and degree of improvement. All acupoints where pharmacopuncture is administered will be recorded at the time of treatment.
  The type and dosage of pharmacopuncture solution to be used during treatment will be determined entirely based on the clinical judgment of the Korean medicine practitioner performing the pharmacopuncture. Retrospective chart reviews will be conducted to record the type of pharmacopuncture solution used and the total amount administered (in ml).
  The treatment will be administered twice a week for a total of 3 weeks, and all sessions will be documented for accurate evaluation.
  Arms: Pharmacopuncture
Procedure: Physical therapy — The selection of physical therapy methods, treatment areas, and treatment duration will be determined based on the clinical judgment of the physician, considering the patient's symptoms, imaging results, and degree of improvement. The type, frequency, and areas of prescribed and administered physical therapy will be recorded.
  The treatment will be administered twice a week for a total of 3 weeks, and all sessions will be documented for accurate evaluation.
  Arms: Physical therapy

SUMMARY:
This study is a pragmatic randomized controlled trial. Condition/disease: Chronic Knee Pain. Intervention: Pharmacopuncture

DETAILED DESCRIPTION:
Knee pain can have various causes. It may result from tears and injuries to structures or from inflammation due to various diseases. Chronic pain is often caused by overuse injuries, inflammation, or arthritis. Among these, osteoarthritis (OA) is the most common cause of chronic pain, affecting approximately 10% of Korean adults aged 20 to 89, either currently or in the past. In addition to OA, other conditions such as rheumatoid arthritis, post-traumatic degenerative arthritis, and chondromalacia can also lead to chronic pain. Therefore, it is evident that a significant number of patients suffer from chronic knee pain.

The purpose of this study is to conduct a pragmatic randomized controlled clinical trial involving 40 patients suffering from chronic knee pain. The trial will compare the effects of treatment strategies utilizing pharmacopuncture (20 patients) with those utilizing the standard Western medical treatment of physical therapy (20 patients) to verify the comparative efficacy of pharmacopuncture.

However, in this pragmatic clinical trial, patients will be randomly assigned to either the pharmacopuncture strategy or the physical therapy strategy. The specific methods of physical therapy and pharmacopuncture will not be predetermined but will be administered based on the clinical judgment of physicians and traditional Korean medicine practitioners according to the patient's condition. All applied treatment methods will be retrospectively reviewed through chart review and recorded in the Case Report Form (CRF) for comparison.

ELIGIBILITY:
Inclusion Criteria:

* Patients whose NRS (Numeric Rating Scale) of knee pain is 5 or higher
* Patients whose symptoms persist for more than 3 months
* Patients who are between 19 and 70 years of age
* Patients who, after receiving a detailed explanation of the clinical study and fully understanding it, voluntarily decide to participate and agree in writing to comply with the precautions.

Exclusion Criteria:

* Patients who have been diagnosed with a specific serious disease that may cause knee pain (acute fracture, dislocation, traumatic damage to ligaments and cartilage, etc.)
* If the cause of the pain is caused by a disease other than the knee (tumor, fibromyalgia, rheumatoid arthritis, gout, lumbar disc herniation, etc.)
* Cases that occur due to a traumatic event and require surgical intervention due to suspected acute fracture, dislocation, ligament and cartilage damage
* Patients who diagnosed other chronic diseases (stroke, myocardial infarction, kidney disease, diabetic neuropathy, dementia, epilepsy, etc.) that may interfere with the treatment effect or interpretation of results.
* Patients who are currently taking steroids, immunosuppressants, drugs for mental illness, or other drugs that may affect the results of the study
* Patients who acupuncture treatment is inappropriate or unsafe: Patients with bleeding disorders, those receiving anticoagulant treatment, and patients with severe diabetes at risk of infection.
* Patients who have taken drugs that may affect pain, such as Non-Steroidal Anti-Inflammatory Drugs (NSAIDs), or have received herbal acupuncture or physical therapy within the past week
* Patients who are pregnant, planning to become pregnant, or are breastfeeding
* Patients within 3 months after knee surgery or if knee replacement surgery was performed
* Patients who has been less than 1 month since you finished participating in another clinical study, or if you are planning to participate in another clinical study during the study participation and follow-up period within 6 months from the date of selection
* Patients who difficult to fill out the consent form for research participation
* Other cases where participation in clinical research is difficult in the judgment of the researcher.

Ages: 19 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2022-12-28 (Actual); Primary Completion 2023-07-12 (Actual); Study Completion 2023-11-30 (Actual)

PRIMARY OUTCOMES:
Knee pain numeric rating scale, NRS | Screening day(W-1), Week 1, 2, 3, 4, 6
  Joint pain will be assessed using the NRS. In the NRS, the patient chooses a number from 0 to 10 that best describes how comfortably they can relax (0 being no pain and 10 being the most comfortable they can imagine).

SECONDARY OUTCOMES:
Knee pain visual analogue scale, VAS | Week 1, 2, 3, 4, 6
  It is an evaluation index that records the degree of pain felt by the patient along a 100 mm horizontal line with one end indicating no pain and the other end indicating the most severe pain imaginable. This is one way to determine the patient's pain level, and the patient enters the degree of knee pain over the past week as a point on a line.
Range of motion, ROM | Screening day(W-1), Week 1, 2, 3, 4, 6
  Passive ROM will be measured before and after treatment to evaluate changes before and after treatment. Passive ROM is evaluated by measuring the angle between the subject's lower extremity and an imaginary line drawn vertically from the ground at the maximum range of motion of the subject's knee joint in flexion, extension, left flexion, and right flexion. If measurement is not possible due to pain, it will be recorded as UC.
Korean Western Ontario & McMaster, K-WOMAC | Week 1, 4, 6
  K-WOMAC is a 24-item questionnaire developed to evaluate the degree of disability related to knee pain. Each question is divided into 5 levels and consists of 5 questions in the pain evaluation section, 2 questions in the stiffness evaluation section, and 17 questions in the functional disability evaluation section. The higher the score, the more severe the disability.
Short Form-12 Health Survey version 2, SF-12 v2 | Week 1, 4, 6
  SF-12 v2 is a questionnaire that evaluates health-related quality of life (HRQoL) and consists of 12 questions in 8 areas (physical functioning, role-physical, bodily pain, general health, vitality, social functioning, role-emotional and mental health). It usually takes less than 5 minutes to complete, and higher scores indicate better health-related quality of life. SF-12 is used to evaluate the functional health and well-being of patients and healthy people. Regarding the Korean version of the SF-12, Kim et al. verified the reliability and validity of its use to measure health-related quality of life in 1,000 Koreans.
EuroQol-5 Dimension, EQ-5D-5L | Week 1, 4, 6
  EQ-5D-5L is a method of evaluating health status from various aspects and then indirectly calculating the quality weight of a specific health status using pre-assigned preference scores for each functional level. It is the most widely used among several indirect measurement methods. there is. The EQ-5D-5L consists of 5 questions. Each question includes mobility, self-care, usual activities, pain/discomfort, and anxiety/depression ( Ask about the level of anxiety/depression, etc. Weights are assigned according to the level of each item, and the preference score calculation equation is presented based on these weights and constants.
Patient Global Impression of Change, PGIC | Week 4, 6
  Patient global impression of change (PGIC) is a method that allows patients to subjectively evaluate the degree of improvement in 7 levels: 1, Very Much Improved; 2, Much Improved; 3, Minimally Improved; 4, No Change; 5, Minimally Worse; 6, Much Worse; or 7, Very Much Worse.
Credibility and Expectancy | Screening day(W-1)
  To evaluate participants' expectations of treatment, a 9-point Likert scale is used.
  At the first visit, participants were asked, "How much do you think herbal acupuncture treatment and physical therapy will relieve your symptoms?" A score will be selected as an answer to the question (1 = not at all, 5 = somewhat, and 9 = very much).
Economic evaluation question-Medical costs | Week 1, 2, 3, 4, 6
  To measure cost items, a separately developed questionnaire was used to measure formal/informal medical costs, non-medical costs, time costs, and productivity loss costs. Formal medical costs are the costs incurred in using the services of medical institutions, while unofficial costs such as purchasing health food and medical equipment are informal medical costs. Costs accompanying the use of medical services, such as transportation costs, patient time costs, and nursing care costs, are non-official costs. Applicable to medical expenses. The cost of productivity loss refers to the cost of economic loss resulting from the inability to participate in labor due to the disease itself or premature death due to the disease. To calculate the cost of productivity loss, a survey will be conducted using WPAI (the Work Productivity and Activity Impairment questionnaire), which will be converted into costs and used for cost-utility analysis.
Economic evaluation question-Time cost | Week 2
  To measure cost items, a separately developed questionnaire was used to measure formal/informal medical costs, non-medical costs, time costs, and productivity loss costs. Formal medical costs are the costs incurred in using the services of medical institutions, while unofficial costs such as purchasing health food and medical equipment are informal medical costs. Costs accompanying the use of medical services, such as transportation costs, patient time costs, and nursing care costs, are non-official costs. Applicable to medical expenses. The cost of productivity loss refers to the cost of economic loss resulting from the inability to participate in labor due to the disease itself or premature death due to the disease. To calculate the cost of productivity loss, a survey will be conducted using WPAI (the Work Productivity and Activity Impairment questionnaire), which will be converted into costs and used for cost-utility analysis.
Economic evaluation question-Productivity loss | Week 1, 2, 3, 4, 6
  To measure cost items, a separately developed questionnaire was used to measure formal/informal medical costs, non-medical costs, time costs, and productivity loss costs. Formal medical costs are the costs incurred in using the services of medical institutions, while unofficial costs such as purchasing health food and medical equipment are informal medical costs. Costs accompanying the use of medical services, such as transportation costs, patient time costs, and nursing care costs, are non-official costs. Applicable to medical expenses. The cost of productivity loss refers to the cost of economic loss resulting from the inability to participate in labor due to the disease itself or premature death due to the disease. To calculate the cost of productivity loss, a survey will be conducted using WPAI (the Work Productivity and Activity Impairment questionnaire), which will be converted into costs and used for cost-utility analysis.

CONTACTS AND LOCATIONS:
Overall Officials: Sunah Kim, KMD, Principal Investigator — Daejeon Jaseng Hospital of Korean Medicine
Locations (1):
- Daejeon Jaseng Hospital of Korean Medicine, Daejeon, South Korea

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Jeong MI, Lim JK, Kim YJ, Jeon YS, Kim S, Kim CY, Park YC, Kim EJ, Hong Y, Nam D, Lee YJ, Kim D, Ha IH. Effectiveness and Safety of Pharmacopuncture Therapy Compared to Standard Physical Therapy in Patients with Chronic Knee Pain: A Pilot Study for a Pragmatic Randomized Controlled Trial. Medicina (Kaunas). 2025 Jun 18;61(6):1106. doi: 10.3390/medicina61061106. PMID 40572793